CLINICAL TRIAL: NCT02058732
Title: Therapeutic Imaging Biomarkers for Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator was unable to fulfill his responsibilities.
Sponsor: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00078370
Record Dates: First submitted 2013-11-08; First posted 2014-02-10 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALS patients receivng stem cells (Active Comparator): Amyotrophic lateral sclerosis(ALS)subjects, who will be receiving stem cells, will undergo a brief clinical evaluation and questionnaire that will last approximately 20 to 30 min. Subjects will be asked to undergo magnetic resonance imaging(MRI)scans of the cervical spine and brain that will last approximately 60 minutes.
  Interventions: Other: MRI
- ALS patients not receiving stem cells (Active Comparator): Amyotrophic lateral sclerosis(ALS)patient who will not be receiving stem cells, will have an MRI that lasts approximately 60 minutes. This MRI will be repeated at three different time points. Subjects will have an initial MRI, then another at both 6 and 12 months after the initial magnetic resonance imaging(MRI)scan. Subjects will also complete a clinical examination which will take approximately 30 minutes for each MRI. The follow-up magnetic resonance imaging(MRI)scans done for ALS patients who do not receive stem cells are part of routine clinical studies and therefore subjects will not be billed.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Subjects will have an MRI that lasts approximately 60 minutes at the same time points as during the stem cell study schedule; once before the stem cell surgery, and again at 1, 6, 12, 18, 24, 36, and 48 months after receiving stem cells. This magnetic resonance imaging(MRI)scan will be of the cervical spine and brain.

SUMMARY:
Study the cervical spinal cord and brain over time to assess changes and differences in subjects with amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Investigators will study cervical spinal cord chemical concentrations and cervical spinal cord and brain microstructure in amyotrophic lateral sclerosis(ALS) patients who have had a stem cell transplant compared to ALS patients who have not had a stem cell transplant. Investigators intend to determine cervical spinal cord chemical concentrations and cervical spinal cord and brain microstructure in amyotrophic lateral sclerosis(ALS) patients who have had a stem cell transplant and compare these to corresponding measures in amyotrophic lateral sclerosis(ALS) patients who have not had a stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Subjects with amyotrophic lateral sclerosis -

Exclusion Criteria:

1. Do not have opportunistic central nervous system infection
2. Do not have a history of head injury
3. Do not have cerebrovascular disease
4. Do not have a contraindication for MRI(e.g. cardiac pacemaker, ferromagnetic or metallic implants).
5. Must not be pregnant -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in spinal cord metabolites in treated ALS subjects and nontreated ALS subjects. | 5 years
  1. The longitudinal changes in spinal cord metabolites in amyotrophic lateral sclerosis(ALS) stem cell treated patients will be compared to amyotrophic lateral sclerosis(ALS) non-treated patients using magnetic resonance spectroscopy. Investigators hypothesize that amyotrophic lateral sclerosis(ALS) stem cell treated patients will demonstrate attenuated rates of decline in the levels of N-acetylaspartate(NAA), a measure of neuronal integrity, in the cervical spinal cord than amyotrophic lateral sclerosis(ALS) non-treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Foerster, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No